CLINICAL TRIAL: NCT04397991
Title: Inhaled Furosemide for Transient Tachypnea of Newborn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Mariam Rajab, Principal Investigator, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 18122018
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Respiratory Morbidity
MeSH Terms: interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Furosemide (Experimental): Patients will receive nebulised furosemide
  Interventions: Other: Furosemide
- Placebo (Placebo Comparator): Patients will receive nebulised 0.9% saline
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Furosemide — Patients will receive nebulised furosemide solution 1 mg/kg
  Arms: Furosemide
Other: Placebo — Patients will receive nebulised 0.9% saline
  Arms: Placebo

SUMMARY:
This is a randomized double blind clinical trial in which newborns with suspected Transient tachypnea of the newborn (TTN) will receive either furosemide or normal saline by nebulizer every 6 hours for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with 34+0-39+0 gestational age
* on the first day of life
* with the clinical diagnosis of Transient Tachypnoea
* need for CPAP >6 hours to obtain the oxygen saturation >92%

Exclusion Criteria:

* Systemic infection
* Intubation and mechanical ventilation before Inclusion in the trail
* Malformation and any other disease with disturb of respiratory system

Ages: 1 Day to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with respiratory morbidity | 24 hours
  Neonatal respiratory morbidity will be assessed through oxygen saturation, respiratory rate and duration on Continuous positive airway pressure (CPAP)

SECONDARY OUTCOMES:
Length of hospital stay | 15 days
  Duration of hospital stay in days

CONTACTS AND LOCATIONS:
Overall Officials: Mariam Rajab, MD, Principal Investigator — Makassed General Hospital
Locations (1):
- Makassed General Hospital, Beirut, Lebanon